CLINICAL TRIAL: NCT04494750
Title: Physiology and Residual Ischemia After Percutaneous Coronary Intervention (EArly Discharge After Transradial Stenting of CoronarY Arteries- EASY- PRIPCI)
Brief Title: Physiology and Residual Ischemia After Percutaneous Coronary Intervention
Acronym: EASY-PRIPCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Quebec Heart Institute (Other)
Responsible Party: Principal Investigator, Olivier F. Bertrand, Director of the International Chair of Interventional Cardiology and Transradial Approach, Laval University
Other Study IDs: EASY-PRIPCI
Record Dates: First submitted 2020-07-27; First posted 2020-07-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Ischemic Heart Disease; Angina Pectoris; Chest Pain; Coronary Artery Disease; Coronary Restenosis
Keywords: Coronary Artery Disease; Fractional Flow Reserve (FFR); Coronary physiology; Repeat intervention; diastolic pressure ratio (dPR)
MeSH Terms: conditions — Myocardial Ischemia; Angina Pectoris; Chest Pain; Coronary Artery Disease; Coronary Restenosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite optimal angiographic result after stent implantation, a number of patients will undergo repeat angiography within 1 year of index procedure. EASY-PRIPCI is an observational study evaluating the incidence of abnormal physiology results in patients undergoing repeat angiography after uncomplicated percutaneous intervention (PCI).

DETAILED DESCRIPTION:
Despite successful PCI and complete revascularization, about 25% of patients will present with angina and/or positive exercise testing during follow-up. With recurring or persistent symptoms, a number of those patients will be referred for control angiography. This might create a significant burden for health systems as well as putting patients to undergo further interventions without clear demonstration of ischemia.

Assessing physiology and fractional flow reserve in particular after PCI could represent a further step to determine whether stent implantation and stenosis removal will be effective to relieve subjective and objective signs of ischemia.

Hypothesis:

Resting gradients such as whole cycle Pd/Pa and diastolic dPR and FFR will be abnormal (below ischemic threshold) in > 20% of cases despite optimal stent implantation and angiographic result.

The use of physiology assessment in previously intervened vessels in patients referred for persisting or recurring angina might help operators to decide upon further intervention.

ELIGIBILITY:
Inclusion Criteria:

* Any patient referred for diagnostic angiography and possible PCI within 12 months of uncomplicated PCI with stent implantation.

Exclusion Criteria:

* Unable to understand study design or objectives of study.
* Unable to sign informed consent.
* Evidence of in-stent restenosis or significant untreated coronary lesions (initial incomplete revascularization)
* Inability to comply with the study follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients returning to the Quebec Heart Institute for a diagnostic angiography and possible PCI within 12 months of a previous uncomplicated PCI with stent implantation.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Rate of successful uncomplicated PCI as per coronary physiology ratios | Transprocedural, initial and final values
  Record the minimal values reported for Pd/Pa, dPR and FFR ratios in the distal vessel after uncomplicated PCI and good angiographic result.Comparison between baseline (pre PCI) and final (post PCI) coronary physiology ratios .

SECONDARY OUTCOMES:
Incidence and types of further interventions or imaging techniques | Historical and immediately after the procedure, up to 36 months
  Record the incidence by type of intervention and diagnostic or imaging techniques
Residual symptoms and quality of life after repeat angiography | up to 30 days
  Identify residual symptoms after intervention, and overall immediate quality of life.
Rates of repeat interventions | Historical and immediately after the procedure
  on previously intervened lesions versus PCI on new lesions
Incidence of successful distal positioning of pressurewire | Transprocedural

CONTACTS AND LOCATIONS:
Overall Officials: Olivier F. Bertrand, MD, PhD, Principal Investigator — Laval University
Locations (1):
- IUCPQ - Laval Hospital, Québec, Canada